CLINICAL TRIAL: NCT04612647
Title: Fit Families Program: Fundamental Motor Skill Intervention in Children With Autism Spectrum Disorders and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-1256; A176000 (Other: UW Madison); EDUC/KINESIOLOGY/KINESIO (Other: UW Madison)
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Workshop group (Experimental): Participants in the workshop group will be offered four one-day workshops (3-hours each) covering topics of 1) Sensory Integration, 2) Communication, 3) Aquatic Opportunities, and 4) Physical activity and Sports (during intervention)-[Parents and Children-Workshop Group]. In addition to the workshops, this group and the home-based group will receive information (activity booklets) and physical education (physical activity)-related equipment.
  Interventions: Other: 12-week FMS Intervention; Behavioral: Physical Activities & Activity Booklets
- Home-based group (Experimental): Participants in the home-based group will not participate in the four half-day workshops, but they will receive the same information (activity booklets) and physical activity equipment as the workshop group (during intervention)-[Parents and Children-Home Group].
  Interventions: Behavioral: Physical Activities & Activity Booklets
- wait-listed home-based group (No Intervention): Wait-list home-based group will serve as the control group (during intervention)-[Parents and Children-Control Group]. This group will be instructed to continue their typical routines and activities for the duration of the intervention. They will be asked to attend the pre and posttest, as well as a follow up three weeks and 3 months after the completion of the 12-week period. Immediately following the follow-up test (3 months after the intervention), participants in the wait-list home-based group will be offered the home-based program (e.g., receiving the same intervention protocol and materials (physical education equipment and lesson plans/workbook) following all procedures as described for that group previously.

INTERVENTIONS:
Other: 12-week FMS Intervention — 4 sessions, no more than 3 hours per session covering 1) Sensory Integration, 2) Communication, 3) Aquatic Opportunities, and 4) Physical activity and Sports (during intervention)
  Arms: Workshop group
Behavioral: Physical Activities & Activity Booklets — expected to engage in physical activity at least 3 hours per week
  Arms: Home-based group; Workshop group

SUMMARY:
The investigators aim to identify the effect of a 12-week fundamental motor skills (FMS) (e.g., throwing, catching, running) intervention on the active participation in physical recreation activities and a variety of other factors (child behaviors, communication, and adaptive skills) and to identify patterns, benefits, constraints, and strategies to active participation in physical recreation activities among families of children with autism spectrum disorders (ASD) (pre-post) through in-person or via phone interviews with parents and children with ASD.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of three protocols: 1) Workshop group, 2) Home-based group, and 3) wait-listed home-based group. Participants in all groups will receive an activity booklet and physical education-related activity items (e.g., ball, hoop). The hypothesis is that both the workshop and home-based groups will improve in all measures from pre to post compared to the wait-list control group. The investigators want to determine if the differences in the workshop and home-based groups differ significantly or are equitable in terms of gains in all areas.

Note: Due to COVID-19 for the post-test, instead of parents attending the UW-Facilities, they will be asked to videotape themselves and their children while performing the test of gross motor development (TGMD) activities. For the follow-up test (Fall 2020) we will expect to conduct these in person. However, if the situation due to COVID-19 remains the same, the investigators will ask families to follow the same procedures (videotape themselves and their children).

ELIGIBILITY:
Parents (one per family) and children with ASD ages 4 to 11 will be included (recruited as a dyad).

Inclusion Criteria:

* ASD must be the primary disability of the child
* Children will be considered to have ASD if they score above the clinical cutoff or 15 on both the lifetime and current versions of the SCQ. Diagnostic severity of ASD will not be a factor in recruitment.
* Children must be able to participate in the program activities.
* Children must be ambulatory and able to follow verbal or picture directions with support
* Children with significant communication needs will still be considered for the study
* No age restriction for adults (parents of children with ASD)
* Parents should be ambulatory and not have any restriction to do physical activity

Exclusion Criteria:

* Parents of children with other primary disabilities, or parents who do not have children with ASD will be excluded.
* Participants cannot exhibit aggressive behavior
* Children who are non-ambulatory, or participants (children) with significant behavioral or sensory impairments will also be excluded based on application information, including existing behavior intervention plans and existing school information

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-05-24 (Actual); Study Completion 2020-05-24 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Development as Measured by TGMD-3 | Baseline, 3 week post intervention (15 weeks), 3 months post intervention (24 weeks)
  The Test of Gross Motor Development - second edition (TGMD-3) is a measure of fundamental motor skills. The total possible range of scores is 47-158, where higher scores are indicative of improved gross motor development.
Number of Participants Whose Perceptions Qualitatively Improve as measured via semi-structured interview | baseline (approximately 2 weeks prior to intervention), post intervention (12 weeks), follow up (24 weeks)
  Children will participate in one-on-one semi-structured interviews with the research team to explore their perception regarding communication strategies (between parent and child), patterns of physical recreation, perceived benefits, and constraints.
Fidelity of Intervention reported as Number of Parents who Implements the Intervention as Intended | up to 12 weeks
  Fidelity checklists will be used to determine the fidelity of the intervention. Parents will be asked to email a video of 1-2 lessons per week along with a completed task analysis checklist. Parents will be asked to confirm whether or not each task was completed on the checklist. The research team will complete the same form while viewing the video to ensure whether the parent knows and is implementing the steps intended and if there are fidelity differences between the workshop and home-based group.
Change in Social Communication Questionnaire (SCQ) | baseline (approximately 2 weeks prior to intervention), post intervention (12 weeks)
  The SCQ is a 40-item survey where each question is a 'yes' or 'no' answer. The total possible range of scores is 0-39 (verbal children) or 0-33 (non-verbal children) with higher scores indicative of greater frequency of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Columna, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No